CLINICAL TRIAL: NCT02883270
Title: Effects of Robotic-assisted Gait Training In Non-Ambulatory Patients After Guillain-Barré Syndrome : A Randomized Controlled Trial
Brief Title: Effects of Robotic-assisted Gait Training In Non-Ambulatory Patients After Guillain-Barré Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Junwei Hao (Other)
Responsible Party: Sponsor-Investigator, Junwei Hao, Tianjin Medical University General Hospital, Tianjin Medical University General Hospital
Organization: Tianjin Medical University General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB2016-039-01
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-09

CONDITIONS: GBS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RAGT treatment group (Experimental): Robotic-assisted gait training （RAGT）is an effective alternative to treadmill therapy with partial body weight in intense gait rehabilitation after some neuropathy. The investigators use LokoHelp for training, which is provided to the feet and the patient actively controls the knee and hip joints. The participants of RAGT treatment group receive 30 min conventional rehabilitation and 30 min robotic-assisted gait training daily for 8 weeks.
  Interventions: Device: Robot-assisted Gait Training
- controls (Placebo Comparator): The participants of controls receive 60 min conventional rehabilitation daily for 8 weeks. Interventions included physiotherapy for muscle strengthening, endurance and gait training; occupational therapy to improve activity of daily living (domestic, community tasks).
  Interventions: Other: conventional rehabilitation

INTERVENTIONS:
Device: Robot-assisted Gait Training — Robot-assisted Gait Training is an effective alternative to treadmill therapy with partial body weight in intense gait rehabilitation and provided to the feet and the patient actively controls the knee and hip joints.
  Other Names: LokoHelp
  Arms: RAGT treatment group
Other: conventional rehabilitation — The participants of controls receive 60 min conventional rehabilitation daily for 8 weeks. Interventions included physiotherapy for muscle strengthening, endurance and gait training; occupational therapy to improve activity of daily living (domestic, community tasks).
  Arms: controls

SUMMARY:
This study investigates the effects of Robotic-assisted gait training in non-ambulatory patients after Guillain-Barré syndrome.The participants are randomly divided into two groups.Patients of the treatment group receive robotic-assisted gait training,while the contorls receive conventional rehabilitation.

DETAILED DESCRIPTION:
Guillain-Barré syndrome (GBS) is an acute autoimmune disease of the peripheral nervous system, which may lead to rapidly developing motor deficits, sensory deficits, autonomic dysfunction and respiratory failure. Approximately, 20.3% of patients cannot walk unaided at 4 weeks of symptom onset and 18.0% at 6 months. So, restoration and improvement of independent walk are one of major goals of GBS rehabilitation. For severely affected neurological patients, gait training using conventional therapy is technically difficult due to their motor weakness and balance problems. Robotic-assisted gait training （RAGT）is an effective alternative to treadmill therapy with partial body weight in intense gait rehabilitation after some neuropathy. And the proven reliability and safety of RAGT suggest that it may be effective for treating non-ambulatory patients after some neuropathy. In our study, we investigated the anti-inflammatory effects of RAGT in non-ambulatory patients of GBS.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of GBS;
* Age between 18 and 65 years;
* Period of GBS is between 4 and 8 weeks;
* severe walking disabilities, defined as a GBS disability score of 2-4;

Exclusion Criteria:

* An unstable phase of disease;
* Disorders preventing RAGT(eg, unstable cardiovascular, respiratory disease ,orthopedic, or neurological condition, unhealed decubitus, orthostatic hypotension etc.) ;
* Severe cognitive impairment preventing meaningful communication;
* Body weight more than 100 kg;
* Pregnancy;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-08; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
GBS disability score | 8 weeks
  0:A healthy state.1:Minor symptoms and capable of running.2:Able to walk 10 m or more without assistance but unable to run.3:Able to walk 10 m across an open space with help.4:Bedridden or chairbound.5:Requiring assisted ventilation for at least part of the day.6:Dead.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No